CLINICAL TRIAL: NCT03033732
Title: Optimizing Patient Centered-Care: A Pragmatic Randomized Control Trial Comparing Models of Care in the Management of Prescription Opioid Misuse (OPTIMA Trial)
Brief Title: A Pragmatic Randomized Control Trial Comparing Models of Care in the Management of Prescription Opioid Misuse
Acronym: OPTIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Didier Jutras Aswad (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Didier Jutras Aswad, Dr. Didier Jutras Aswad - Principal Investigator, Canadian Research Initiative in Substance Misuse
Organization: Canadian Research Initiative in Substance Misuse (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRISM 001
Record Dates: First submitted 2017-01-10; First posted 2017-01-27 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Opioid Use Disorder
Keywords: opioid agonist treatment; pragmatic; prescription opioid use; patient engagement
MeSH Terms: conditions — Opioid-Related Disorders; Patient Participation | interventions — Methadone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Other): Opioid agonist treatment for opioid use disorder. Ingested in liquid oral form via strict initial daily witnessed ingestion as per local guidelines.
  Interventions: Drug: Methadone
- Buprenorphine/Naloxone (Other): Opioid agonist treatment for opioid use disorder. Ingested orally via sublingual tablet form, flexible take home dosing.
  Interventions: Drug: Buprenorphine-Naloxone

INTERVENTIONS:
Drug: Methadone — Methadone is a synthetic analgesic drug used as a substitute drug in the treatment of opioid use disorder. Methadone is administered via strict daily witnessed ingestion.
  Other Names: Methadose
  Arms: Methadone
Drug: Buprenorphine-Naloxone — Buprenorphine/Naloxone is an opioid agonist treatment used to treat opioid use disorder. Buprenorphine/Naloxone is administered via flexible take home dosing once the patient has reached stabilization as per physician discretion.
  Other Names: Suboxone
  Arms: Buprenorphine/Naloxone

SUMMARY:
This trial evaluates two standard of care treatments for opioid addiction: methadone and buprenorphine/naloxone. In order to improve patient care, the study will address real-world treatment conditions, including strict regulations for methadone dosing (i.e. initially dispensed daily at the pharmacy until stabilisation) vs. flexible take-home dosing for buprenorphine/naloxone. The OPTIMA study is designed with the intention to support patient-provider decision-making and evaluate health related outcomes with the overall aim of improving treatment outcomes through enhancing patient-centered approaches in clinical care.

DETAILED DESCRIPTION:
This is a multicenter, open-label, 2-arm, randomized trial with a pragmatic design involving 276 individuals with prescription opioid use disorder. Participants will be randomized to receive either:

1. Methadone provided via initial daily witnessed ingestion as per local guidelines.
2. Buprenorphine/naloxone maintenance therapy provided via flexible take-home dose regimens dispensed as per the physician's discretion, once clinical stability is achieved.

Once randomized to a study medication and treatment initiation and induction has begun, study physicians and participants will discuss the treatment plans and procedures going forward. Once treatment initiation has taken place, the participant will attend study visits every 2 weeks (including collection of urine samples) for the 24-week intervention period. For all study sites, standardized guidelines exist and will be adhered to for the safe induction of both medications. Frequency of illicit opioid use, intensity of craving and other secondary endpoints will also be assessed via standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged between 18 and 64 years of age inclusively;
2. Prescription opioid use disorder (as defined by the Diagnostic and Statistical Manual of Mental Disorders-5 criteria), which requires opioid agonist therapy as per the discretion of the physician;
3. Female participants may be eligible if:

   1. Is of non-childbearing potential, defined as (i) post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age); or (ii) documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy).
   2. Is of childbearing potential, has a negative pregnancy test at screening and and agrees to use an acceptable method of birth control throughout study;
4. Be willing to be randomized to 24 weeks of either methadone or buprenorphine/naloxone adapted model of care, and to be followed for the duration of the trial;
5. Be able to provide written informed consent;
6. Be willing to comply with study procedures;
7. Be able to communicate in English or French.

Exclusion Criteria:

1. Any disabling medical condition as assessed by medical history, physical exam, vital signs and/or laboratory assessments that, in the opinion of the study physician, precludes the safe participation in the study or the ability to provide fully informed consent;
2. Any disabling, unstable or acute mental condition that in the opinion of the study physician precludes safe participation in the study or ability to provide fully informed consent;
3. Heroin reported as the most frequently used opioid in the past 30 days;
4. Taken methadone or buprenorphine/naloxone for Opioid Use Disorder maintenance treatment in the four weeks prior to screening;
5. Pain of sufficient severity as to require ongoing pain management with opioids;
6. History of a severe adverse event, hypersensitivity reaction, or allergic reaction to either methadone or buprenorphine/naloxone;
7. Pregnant, nursing, or planning to become pregnant during the study period;
8. Currently taking or have taken an investigational drug in another study in the last 30 days, confirmed via self-report;
9. Pending legal action or other reasons in the opinion of the study physician that might prevent completion of the study;
10. Presence of a substance use disorder that, in the opinion of the study physician, precludes safe participation in the study (e.g. unstable or severe alcohol use disorder, unstable or severe benzodiazepine use disorder);
11. Current treatment with medications that may interact with either methadone or buprenorphine/naloxone (e.g. Clonazepam, Benzodiazepines) OR anticipation that the patient may need to initiate such treatment during the trial that is deemed unsafe by the study physician or could prevent study completion;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Opioid Use | 24 weeks
  Opioid use will be measured by the overall proportion of opioid-free urine drug screens (UDS) during the 24 weeks of the trial (excluding the assigned metabolites of opioid agonist treatments, as appropriate), with missing values defined as positive UDS (binary, laboratory assay).

SECONDARY OUTCOMES:
Retention in treatment | 24 weeks
  Retention in treatment is defined as the proportion of participants on assigned opioid agonist treatment (OAT) at the end of the study, as defined by having both a) an active prescription for the assigned OAT at week 24, and b) a positive UDS result for the assigned OAT at week 24.
Opioid Agonist Treatment (OAT) Medication Adherence | 24 weeks
  OAT medication adherence is defined as the proportion of assigned treatment doses received over the 24-week trial period assessed by both Pharmacy Abstraction and participant self-report.
Safety will be evaluated by monitoring adverse events (AEs) and serious adverse events (SAEs) | 24 weeks
  Safety will be evaluated by monitoring adverse events (AEs) and serious adverse events (SAEs) throughout the duration of the trial. Adverse events and SAEs will be collected during study visits by means of open questions (e.g., has there been any changes to your health since the last study visit?). Also, the observation of clinically significant change in lab test results, fatal or non-fatal overdoses, and precipitated withdrawal symptoms from buprenorphine/naloxone inductions will be used to document AEs and SAEs. All AEs and SAEs will be documented using an AE Log in which the date and time of onset, the end date and time (i.e., when the AE was resolved or stabilized), the severity of the event, any action taken with respect to the study medication (e.g., no treatment or dose adjustment), and the relationship with study protocol or study medication will be recorded.
Patient Satisfaction | 24 weeks
  Patient satisfaction to the assigned treatment will be recorded on the Client Satisfaction Questionnaire (CSQ-8) and will be administered at 4, 12, and 24 weeks (end of study).
Patient Engagement | 24 weeks
  Patient engagement in treatment will be measured through self-report questionnaires administered at Treatment Initiation, week 4, week 12, and week 24 visits. The primary measure of ongoing patient engagement will be administered at Treatment Initiation and every 2 weeks.

OTHER OUTCOMES:
Quality of life | 24 weeks
  Quality of Life (QoL) will be evaluated via the EQ5-D self-report questionnaires administered at Treatment Initiation and every 4 weeks.
Pain | 24 weeks
  Pain will be assessed via Brief Pain Inventory self-report questionnaire at Screening to determine eligibility, Treatment Initiation and every 4 weeks for the 24 week intervention period.
Proportion of Participants who Initiate Taper | 24 weeks
  The proportion of patients who initiate taper will be assessed by using a standardized induction case report form completed via both pharmacy abstraction and self-report. The pharmacy record abstraction will collect information on opioid agonist treatment use and on the days between follow up visits, as well as information on end or switching of opioid agonist treatments, missing doses and reason any change in medication status or dose change. The participant will also be asked about his/her use of opioid agonist treatments in the past 2 weeks or since the last study visit collecting information similar to that information collected in the pharmacy abstraction.
Cost-effectiveness | 24 weeks
  Information on health service utilization will be collected at baseline and every 4 weeks for the 24-week intervention period. Items were selected from modules selected from the European Addiction Severity Index which collect self-report data on income, medical/medication status, healthcare provider visits, and criminal activity. This information will either be collected on paper source or entered by the participant directly into the Electronic Data Capture (EDC) system.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras Aswad, MD, Principal Investigator — Canadian Research Initiative in Substance Misuse; Maria E Socias, MD, Principal Investigator — British Columbia Centre on Substance Use; Keith Ahamad, MD, Principal Investigator — British Columbia Centre on Substance use; Bernard LeFoll, PhD, Principal Investigator — Centre for Addiction and Mental Health; Ron Lim, MD, Principal Investigator — University of Calgary; Julie Bruneau, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Evan Wood, MD, Principal Investigator — British Columbia Centre on Substance Use; Cameron Wild, PhD, Principal Investigator — University of Alberta; Jurgen Rehm, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (7):
- Canada (7):
  - Calgary Opioid Dependency Program, Calgary, Alberta
  - Edmonton Opioid Dependency Program, Edmonton, Alberta
  - Rapid Access Addictions Clinic-St. Paul's Hospital, Vancouver, British Columbia
  - Ontario Addiction Treatment Centres- Sudbury Clinic, Greater Sudbury, Ontario
  - Addiction Medicine Service- Centre for Addictions and Mental Health, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Centre de Recherche et d'Aide pour Narcomane, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bastien G, Abboud A, McAnulty C, Mahroug A, Le Foll B, Socias ME, Juteau LC, Dubreucq S, Jutras-Aswad D. Concordance Between Urine Drug Screening and Self-Reported Use in the Context of a Pragmatic Randomized-Controlled Trial in People with Prescription-Type Opioid Use Disorder: Concordance entre le depistage de drogues dans l'urine et l'usage autodeclare dans le contexte d'un essai pragmatique controle a repartition aleatoire chez des personnes presentant un trouble lie a l'usage d'opioides vendus sur ordonnance. Can J Psychiatry. 2026 Jan;71(1):41-52. doi: 10.1177/07067437251367180. Epub 2025 Aug 28. PMID 40874578
- [Derived] Bouthillier A, Bastien G, McAnulty C, Bakouni H, Le Foll B, Socias ME, Jutras-Aswad D. Opioid consumption frequency and its associations with potential life problems during opioid agonist treatment in individuals with prescription-type opioid use disorder: exploratory results from the OPTIMA Study. Harm Reduct J. 2025 Feb 8;22(1):14. doi: 10.1186/s12954-025-01157-4. PMID 39923043
- [Derived] Langlois J, Fairbairn N, Jutras-Aswad D, Le Foll B, Lim R, Socias ME. Characterising methamphetamine/amphetamine use among opioid agonist therapy-seeking adults with prescription-type opioid use disorder in Canada. Drug Alcohol Rev. 2024 Nov;43(7):1905-1912. doi: 10.1111/dar.13863. Epub 2024 May 9. PMID 38721650
- [Derived] Bastien G, Abboud A, McAnulty C, Elkrief L, Ledjiar O, Socias ME, Le Foll B, Bahji A, Brissette S, Marsan S, Jutras-Aswad D. Impact of Depressive Symptom Severity on Buprenorphine/Naloxone and Methadone Outcomes in People With Prescription-Type Opioid Use Disorder: Results From a Pragmatic Randomized Controlled Trial. J Dual Diagn. 2024 Jul-Sep;20(3):189-200. doi: 10.1080/15504263.2024.2329267. Epub 2024 Apr 5. PMID 38580298
- [Derived] Socias ME, Cui Z, Le Foll B, Lei J, Stewart S, Anand R, Jutras-Aswad D. Sexually transmitted and blood-borne infection risk reduction with methadone and buprenorphine/naloxone among people with prescription-type opioid use disorder: Findings from a Canadian pragmatic randomized trial. HIV Med. 2024 Jul;25(7):817-825. doi: 10.1111/hiv.13636. Epub 2024 Mar 20. PMID 38506171
- [Derived] Bahji A, Bastien G, Bach P, Choi J, Le Foll B, Lim R, Jutras-Aswad D, Socias ME. The Association Between Self-Reported Anxiety and Retention in Opioid Agonist Therapy: Findings From a Canadian Pragmatic Trial. Can J Psychiatry. 2024 Mar;69(3):172-182. doi: 10.1177/07067437231194385. Epub 2023 Sep 12. PMID 37697811
- [Derived] Elkrief L, Bastien G, McAnulty C, Bakouni H, Hebert FO, Socias ME, Le Foll B, Lim R, Ledjiar O, Marsan S, Brissette S, Jutras-Aswad D; OPTIMA Research Group within the Canadian Research Initiative in Substance Misuse. Differential effect of cannabis use on opioid agonist treatment outcomes: Exploratory analyses from the OPTIMA study. J Subst Use Addict Treat. 2023 Jun;149:209031. doi: 10.1016/j.josat.2023.209031. Epub 2023 Mar 30. PMID 37003540
- [Derived] Bastien G, McAnulty C, Ledjiar O, Socias ME, Le Foll B, Lim R, Hassan AN, Brissette S, Marsan S, Talbot A, Jutras-Aswad D; OPTIMA Research Group within the Canadian Research Initiative in Substance Misuse. Effects of Buprenorphine/Naloxone and Methadone on Depressive Symptoms in People with Prescription Opioid Use Disorder: A Pragmatic Randomised Controlled Trial. Can J Psychiatry. 2023 Aug;68(8):572-585. doi: 10.1177/07067437221145013. Epub 2022 Dec 14. PMID 36519188
- [Derived] McAnulty C, Bastien G, Eugenia Socias M, Bruneau J, Le Foll B, Lim R, Brissette S, Ledjiar O, Marsan S, Talbot A, Jutras-Aswad D; OPTIMA Research Group within the Canadian Research Initiative in Substance Misuse. Buprenorphine/naloxone and methadone effectiveness for reducing craving in individuals with prescription opioid use disorder: Exploratory results from an open-label, pragmatic randomized controlled trial. Drug Alcohol Depend. 2022 Oct 1;239:109604. doi: 10.1016/j.drugalcdep.2022.109604. Epub 2022 Aug 17. PMID 36037586
- [Derived] Jutras-Aswad D, Le Foll B, Ahamad K, Lim R, Bruneau J, Fischer B, Rehm J, Wild TC, Wood E, Brissette S, Gagnon L, Fikowski J, Ledjiar O, Masse B, Socias ME; OPTIMA Research Group within the Canadian Research Initiative in Substance Misuse. Flexible Buprenorphine/Naloxone Model of Care for Reducing Opioid Use in Individuals With Prescription-Type Opioid Use Disorder: An Open-Label, Pragmatic, Noninferiority Randomized Controlled Trial. Am J Psychiatry. 2022 Oct;179(10):726-739. doi: 10.1176/appi.ajp.21090964. Epub 2022 Jun 15. PMID 35702828
- [Derived] Socias ME, Ahamad K, Le Foll B, Lim R, Bruneau J, Fischer B, Wild TC, Wood E, Jutras-Aswad D. The OPTIMA study, buprenorphine/naloxone and methadone models of care for the treatment of prescription opioid use disorder: Study design and rationale. Contemp Clin Trials. 2018 Jun;69:21-27. doi: 10.1016/j.cct.2018.04.001. Epub 2018 Apr 5. PMID 29627621